CLINICAL TRIAL: NCT07363733
Title: Randomized Clinical Trial of the Efficacy of Combined Dynamic Quadripolar Radiofrequency Therapy VS Topical Corticosteroid Therapy in Women With Vulvar Lichen Sclerosus
Brief Title: Dynamic Quadripolar Radiofrequency VS Topical Corticosteroids in Women With Vulvar Lichen Sclerosus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal State Budget Institution Research Center for Obstetrics, Gynecology and Perinatology Ministry of Healthcare (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DQRF10.2025
Record Dates: First submitted 2025-12-28; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Vulvar Lichen Sclerosus
Keywords: vulvar lichen sclerosus; Dynamic Quadripolar RadioFrequency; Glucocorticoids; Immunohistochemistry; Quality of Life; Female Sexual Function
MeSH Terms: conditions — Vulvar Lichen Sclerosus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic Quadripolar Radiofrequency Plus Topical Corticosteroids (Experimental): Participants receive topical high-potency corticosteroid therapy according to the standardized regimen, followed by combined Dynamic Quadripolar Radiofrequency (DQRF) therapy initiated 2 weeks after the start of corticosteroid treatment.
  Interventions: Device: Dynamic Quadripolar Radiofrequency (DQRF); Drug: Topical high-potency corticosteroid
- Topical Corticosteroid Monotherapy (Active Comparator): Participants receive topical high-potency corticosteroid therapy according to a standardized treatment regimen.
  Interventions: Drug: Topical high-potency corticosteroid

INTERVENTIONS:
Device: Dynamic Quadripolar Radiofrequency (DQRF) — Dynamic quadripolar radiofrequency therapy administered according to a standardized treatment protocol consisting of four sessions performed at two-week intervals.
  Arms: Dynamic Quadripolar Radiofrequency Plus Topical Corticosteroids
Drug: Topical high-potency corticosteroid — Topical high-potency corticosteroid therapy administered according to the same standardized treatment regimen as in the control arm.

SUMMARY:
This is a prospective, randomized study in women of reproductive age with vulvar lichen sclerosus. Participants will be randomly assigned by investigators using a computer-generated sequence to receive either combined dynamic quadripolar radiofrequency (DQRF) plus topical corticosteroid therapy or topical high-potency corticosteroid therapy alone. Clinical outcomes, patient-reported outcomes and tissue-level changes evaluated by histology, elastin histochemistry, and immunohistochemistry for estrogen, androgen receptors and superoxide dismutase 2 (SOD2) will be assessed before and after treatment, and during follow-up at 3, 6, and 12 months. Safety will be monitored throughout the study. Histochemical and immunohistochemical analyses will be performed in a subset of 10 patients per group before the treatment and at 3 months after the completion of treatment.

DETAILED DESCRIPTION:
This is a prospective, randomized study conducted in women reproductive age with vulvar lichen sclerosus. Computer-generated randomization using an electronic spreadsheet will be used by investigators to assign participants to study groups.

Study groups Group 1: topical high-potency corticosteroid therapy according to the standardized regimen, followed by combined Dynamic Quadripolar Radiofrequency (DQRF) therapy initiated 2 weeks after the start of corticosteroid treatment. DQRF therapy will be administered using a small vulvar applicator in a total of four sessions, performed at two-week intervals.

Group 2: topical high-potency corticosteroid therapy according to a standardized regimen.

Study assessments Clinical assessment At baseline and each follow-up visit, participants will undergo standardized vulvar examination with documentation of objective signs (skin color changes, sclerosis, fissures, erosions, scarring and architectural changes) and symptom severity. Clinical severity will be assessed using a structured clinician-rated vulvar lichen sclerosus severity score. Standardized photo documentation will be performed.

Patient-reported outcome measures

Patient-reported outcomes will be assessed using validated questionnaires:

* Numeric Rating Scale (NRS) for pruritus, vulvar pain, burning, dryness and dyspareunia;
* Vulvar Quality of Life Index (VQLI);
* Short Form-12 Health Survey (SF-12);
* Female Sexual Function Index (FSFI). Histological and tissue-level assessment

Histochemical and immunohistochemical analyses will be performed in a subset of 10 patients per group. Vulvar punch biopsy specimens will be obtained before initiation of therapy and after completion of treatment for:

* immunohistochemical analysis of estrogen receptors, androgen receptors and superoxide dismutase 2 (SOD2) expression;
* histochemical assessment of elastin fiber staining intensity and distribution using a standardized elastin stain, with semi-quantitative grading and/or digital image analysis.

Safety assessment Adverse events related to topical therapy, radiofrequency treatment will be recorded throughout the study.

Follow-up period Participants will be followed longitudinally before the treatment, at the end of treatment, and at 3, 6, and 12 months after completion of therapy to evaluate short-term response, durability of clinical improvement, and disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 49 years (women of reproductive age);
* Histologically confirmed diagnosis of vulvar lichen sclerosus;
* Written informed consent to participate in the study.

Exclusion Criteria:

* Pregnancy or lactation;
* Malignancy at the time of treatment or during any period of follow-up;
* Postmenopausal status;
* Severe decompensated somatic disease;
* Sexually transmitted infections, including hepatitis B, hepatitis C, and syphilis;
* Presence of a cardiac pacemaker or metal-containing intrauterine device (IUD);
* History of treatment with other high-energy-based modalities within the last 6 months;
* Use of topical corticosteroids within the last 3 months;
* Immunosuppression, including immunodeficiency disorders (such as HIV/AIDS) or use of immunosuppressive medications;
* Psychiatric disorders or communication difficulties that may interfere with study participation or compliance.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in clinical severity of vulvar lichen sclerosus | Before treatment (baseline), at the end of treatment, and at 3, 6, and 12 months after completion of therapy.
  Change from baseline in patient-reported symptom intensity using validated questionnaire (Numeric Rating Scale (NRS) for pruritus, vulvar pain, burning, dryness and dyspareunia).

SECONDARY OUTCOMES:
Changes in Patient-Reported Outcomes | Before treatment (baseline), at the end of treatment, and at 3, 6, and 12 months after completion of therapy.
  Change from baseline in general health-related quality of life assessed using the Short Form-12 Health Survey (SF-12). Change from baseline in sexual function assessed using the Female Sexual Function Index (FSFI).
Tissue-Level Biomarkers | Before treatment (baseline) and at 3 months after completion of therapy.
  Change from baseline in estrogen and androgen receptor expression (percentage) in vulvar tissue assessed by immunohistochemistry in a subset of 10 patients per group. Change from baseline in superoxide dismutase (SOD) expression (percentage) in vulvar tissue assessed by immunohistochemistry in a subset of 10 patients per group. Change from baseline in elastin fiber staining intensity (percentage) and distribution in vulvar tissue assessed by histochemical analysis in a subset of 10 patients per group.

CONTACTS AND LOCATIONS:
Overall Officials: Khava Balashova, MD, Obstetrics and Gynecology, Principal Investigator — National Medical Research Center for Obstetrics, Gynecology and Perinatology named after Academician V.I. Kulakov, Ministry of Health of the Russian Federation
Locations (1):
- National Medical Research Center for Obstetrics, Gynecology and Perinatology named after Academician V.I. Kulakov, Ministry of Health of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
Patients data is available upon request from the authors with no identifiable information